CLINICAL TRIAL: NCT06390059
Title: PANOVA-4: Pilot, Single Arm Study of Tumor Treating Fields (TTFields, 150kHz) Concomitant With Atezolizumab, Gemcitabine and Nab-Paclitaxel as First-Line Treatment for Metastatic Pancreatic Ductal Adenocarcinoma (mPDAC)
Brief Title: EF-39 PANOVA-4: Study of Tumor Treating Fields Concomitant With Atezolizumab, Gemcitabine and Nab-Paclitaxel as First-LineTreatment for Metastatic Pancreatic Ductal Adenocarcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EF-39; EF-39 (Other: Sponsor); 2022-003157-55 (EudraCT Number)
Record Dates: First submitted 2024-02-29; First posted 2024-04-29 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Pancreatic Ductal Adenocarcinoma
Keywords: EF-39; PANOVA-4; metastatic pancreatic cancer; tumor treating fields; atezolizumab; gemcitabine and nab-paclitaxel; first line treatment; mPDAC
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — atezolizumab; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, single arm, multi-center, historical control pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TTFields + atezolizumab + gemcitabine and nab-paclitaxel (Experimental): Patients receive TTFields at 150 kHzconcomitant with atezolizumab, gemcitabine and nab-paclitaxel until disease progression or loss of clinical benefit.
  Interventions: Device: Tumor Treating Fields; Drug: Atezolizumab; Drug: Gemcitabine; Drug: nab-paclitaxel

INTERVENTIONS:
Device: Tumor Treating Fields — The NovoTTF-200T is a portable, battery operated system intended for continuous home use, which delivers TTFields at a frequency of 150kHz to the patient by means of insulated transducer arrays. The NovoTTF-200T produces TTFields that exert electric forces intended to disrupt cancer cell division.
  TTFields at 150 kHz application will be continuous for at least 18 hours a day on average. TTFields will be continued until disease progression according to RECISTv1.1 or loss of clinical benefit.
  Other Names: NovoTTF-200T
Drug: Atezolizumab — Atezolizumab is a humanized IgG1 monoclonal antibody which targets human PD-L1and inhibits its interaction with its receptors, PD-1 and B7.1 (CD80). Both of these interactions are reported to provide inhibitory signals to T cells. Atezolizumab is administered as an intravenous solution.
  Atezolizumab may continue until disease progression according to RECIST v1.1 or loss of clinical benefit.
  Other Names: Tecentriq (Brand name)
Drug: Gemcitabine — Gemcitabine is a standard of care chemotherapy drug administered as an intravenous infusion.
  Gemcitabine may continue until disease progression according to RECIST v1.1 or loss of clinical benefit.
  Other Names: Gemzar
Drug: nab-paclitaxel — Nab-paclitaxel is a standard of care chemotherapy drug administered as an intravenous infusion.
  Nab-paclitaxel may continue until disease progression according to RECIST v1.1 or loss of clinical benefit.
  Other Names: Abraxane

SUMMARY:
The PANOVA-4 study is designed to evaluate the safety and efficacy of Tumor Treating Fields (TTFields) therapy together with atezolizumab, gemcitabine and nab-paclitaxel, for the treatment of metastatic pancreatic cancer. The study is intended for patients who have been diagnosed with metastatic pancreatic cancer and have not received prior systemic therapy.

DETAILED DESCRIPTION:
The PANOVA-4 study is an international, multi-center, research study for female and male adult patients diagnosed with metastatic pancreatic ductal adenocarcinoma (mPDAC).

The purpose of the study is to test the efficacy and safety of TTFields, delivered using the NovoTTF-200T Treatment Kit, concomitantly with atezolizumab, gemcitabine and nab-paclitaxel as first line treatment for Metastatic Pancreatic Ductal Adenocarcinoma (mPDAC).

The chemotherapy used in this study, gemcitabine and nab-paclitaxel, are standard-of-care treatment for metastatic pancreatic cancer. The atezolizumab drug and the NovoTTF-200T device are investigational for this tumor type. Atezolizumab is an immunotherapy drug that works with the immune system to help fight cancer. NovoTTF-200T is a non-invasive medical device that delivers Tumor Treating Fields (TTFields) at 150kHz to the cancer in the abdominal region, where the tumor is located.

The study is expected to enroll 76 patients in centers around the world. The expected duration on study per patient is approximately 12 months.

Patients with previously untreated mPDAC who meet all inclusion criteria and none of the exclusion criteria as determined by the investigator will initiate study treatment within 28 days from signing the Informed Consent Form (ICF) to receive TTFields (150 kHz), atezolizumab, gemcitabine and nab-paclitaxel.

All patients enrolled in the study will receive continuous TTFields therapy concomitant with monthly atezolizumab treatments for their metastatic pancreatic cancer and weekly gemcitabine and nab-paclitaxel.

While on the study, patients will be asked to visit the clinic every 4 weeks, in order to perform a physical examination, blood tests,and some other assessments. Patients will be asked to have a radiological examination (CT scan of the chest abdomen and pelvis) every 8 weeks to assess the status of the disease.

Study treatments will continue until disease progression according to RECIST v1.1, or loss of clinical benefit.

Patients who experience disease progression will be permitted to continue study treatments if there is evidence of clinical benefit.

Subjects will return to the clinic for one final visit approximately 30 days after discontinuation of the last study treatment.

Following the final visit, the subjects will be contacted every three months by telephone to answer basic questions about their health status.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form for the study protocol.
2. 18 years of age and older at the time of signing Informed Consent Form.
3. ECOG (Eastern Cooperative Oncology Group) performance status of 0-1.
4. Histologically or cytologically confirmed de-novo diagnosis of metastatic pancreatic ductal adenocarcinoma (PDAC).
5. No prior treatment for PDAC.
6. Life expectancy equal to or greater than 3 months.
7. Measurable disease in the abdomen, as defined by RECIST (Response Evaluation Criteria in Solid Tumors) v1.1.
8. Preferably, tumor accessible for tissue collection. Consent to provide blood and tumor tissue for exploratory study is highly encouraged. Patients who cannot or are unwilling to provide tissue or blood for the exploratory study are not excluded from the study.

   * If tumor tissue is available, a formalin-fixed, paraffin-embedded (FFPE) tumor specimen in a paraffin block (preferred) or approximately 10-15 slides containing unstained, freshly cut, serial sections should be submitted along with an associated pathology report prior to study treatment initiation.
   * If FFPE specimens described above are not available, any type of specimens (including fine-needle aspiration, cell pellet specimens [e.g., from pleural effusion], and lavage samples) are also acceptable. This specimen should be accompanied by the associated pathology report.
   * As mentioned above, if tumor tissue is not available (e.g., depleted because of prior diagnostic testing), patients are still eligible.
9. Amenable and assigned by the investigator to receive therapy with gemcitabine and nab- paclitaxel.
10. Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 14 days prior to initiation of study treatment:

    1. ANC (absolute neutrophil count) ≥ 1.5 X 109/L (1500/μL) without granulocyte colony-stimulating factor support within 14 days prior to initiation of study treatment.
    2. Lymphocyte count ≥ 0.5 X 109/L (500/μL).
    3. WBC (white blood cell) count ≥2.5x109/L (2500/ μL).
    4. Platelet count ≥ 100 X 109/L (100,000/μL) without transfusion.
    5. Hemoglobin ≥ 90 g/L (9 g/dL). Patients may be transfused to meet this criterion.
    6. AST (aspartate aminotransferase), ALT (alanine aminotransferase), and ALP (alkaline phosphatase) ≤ 2.5 X upper limit of normal (ULN), with the following exceptions:

       • Patients with documented liver metastases: AST and/or ALT ≤ 5 X ULN. Patients with documented liver or bone metastases: ALP ≤ 5 X ULN.
    7. Total bilirubin ≤ 1.5 X ULN with the following exception:

       • Patients with known Gilbert disease: total bilirubin ≤ 3 X ULN.
    8. Creatinine ≤ 1.5 X ULN.
    9. Albumin ≥ 25 g/L (2.5 g/dL).
    10. For patients not receiving therapeutic anticoagulation: INR/PT (international normalized ratio/ prothrombin time) or aPTT/PTT (activated partial thromboplastin time/partial thromboplastin time) ≤ 1.5 X ULN.
11. For patients receiving therapeutic anticoagulation: stable anticoagulation regimen.
12. Negative hepatitis B surface antigen (HBsAg) test at screening
13. Positive hepatitis B surface antibody (HBsAb) test at screening, or negative HBsAb at screening accompanied by either of the following:

    * Negative total hepatitis B core antibody (HBcAb)
    * Positive total HBcAb test followed by a negative (per local laboratory definition) hepatitis B virus (HBV) DNA (deoxyribonucleic acid) test. The HBV DNA test must be performed for patients who have a negative HBsAg test, a negative HBsAb test, and a positive total HBcAb test.
14. Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA (Ribonucleic acid) test at screening The HCV RNA test must be performed for patients who have a positive HCV antibody test.
15. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception and agreement to refrain from donating eggs, as defined below:

    * Women must remain abstinent or use contraceptive methods with a failure rate of <1% per year during the treatment period, for 5 months after the final dose of atezolizumab, for 6 months after the final dose of gemcitabine and for 6 months after the final dose of nab-paclitaxel. Women must refrain from donating eggs during this same period.
    * A woman is considered to be of childbearing potential if she is post-menarchal, has not reached a postmenopausal state (≥12 continuous months of amenorrhea with no identified cause other than menopause),and is not permanently infertile due to surgery (i.e. removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the investigator (e.g., Müllerian agenesis). The definition of childbearing potential may be adapted for alignment with local guidelines or regulations.
    * Examples of contraceptive methods with a failure rate of <1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptive that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
    * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not adequate methods of contraception. If required per local guidelines or regulations, locally recognized adequate methods of contraception and information about the reliability of abstinence will be described in the local Informed Consent Form.
    * All patients who are capable of becoming pregnant must take a pregnancy test which is negative within 72 hours before initiation of study treatment.
16. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agreement to refrain from donating sperm, as defined below:

    With a female partner of childbearing potential who is not pregnant, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of <1% per year during the treatment period and for 6 months after the final dose of gemcitabine and for 6 months after the final dose of nab-paclitaxel. Men must refrain from donating sperm during this same period.

    With a pregnant female partner, men must remain abstinent or use a condom during the treatment period and for 6 months after the final dose of gemcitabine and for 6 months after the final dose of nab-paclitaxel to avoid exposing the embryo.

    The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not adequate methods of contraception. If required per local guidelines or regulations, locally recognized adequate methods of contraception and information about the reliability of abstinence will be described in the local Informed Consent Form.
17. Able to operate the NovoTTF-200T device independently or with the help of a caregiver.

Exclusion Criteria:

1. Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases.

   Asymptomatic patients with treated CNS lesions are eligible, provided that all of the following criteria are met:
   * The patient has no history of intracranial hemorrhage or spinal cord hemorrhage.
   * The patient has not undergone stereotactic radiotherapy within 7 days prior to initiation of study treatment, whole-brain radiotherapy within 14 days prior to initiation of study treatment, or neurosurgical resection within 28 days prior to initiation of study treatment.
   * The patient has no ongoing requirement for corticosteroids as therapy for CNS disease.
   * Anticonvulsant therapy at a stable dose is permitted.
2. History of leptomeningeal disease.
3. Uncontrolled tumor-related pain

   * Patients requiring pain medication must be on a stable regimen at study entry.
   * Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to treatment initiation. Patients should be recovered from the effects of radiation. There is no required minimum recovery period. Palliative radiotherapy is permitted, provided it does not interfere with the assessment of tumor target lesions (e.g., the lesion to be irradiated must not be the only site of measurable disease).
   * Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for loco-regional therapy, if appropriate, prior to treatment initiation.
4. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring drainage procedure (i.e., more than one time per month).

   • Patients with indwelling catheters (e.g. PleurX®) are allowed
5. Uncontrolled or symptomatic hypercalcemia (ionized calcium >1.5 mmol/L, calcium >12 mg/dL, or corrected calcium>ULN)
6. Active or history of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome or multiple sclerosis (see Appendix 2 for a more comprehensive list of autoimmune diseases and immune deficiencies), with the following exceptions:

   * Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid-replacement hormone may be eligible for this study
   * Patients with controlled Type 1 diabetes mellitus on a stable insulin regimen are eligible for this study
   * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g. patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

     * Rash must cover <10% of body surface area
     * Disease is well controlled at baseline and only requiring low-potency topical steroids
     * No acute exacerbations of underlying condition within the last 12 months requiring treatment with either psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral steroids
7. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan.

   History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
8. Positive human immunodeficiency (HIV) test at screening or at any time prior to screening.
9. Current treatment with anti-viral therapy for HBV (hepatitis B virus).
10. Active tuberculosis.
11. Severe infection within 4 weeks prior to initiation of study treatment, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia, or any active infection that, in the opinion of the investigator, could impact patient safety.
12. Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab.
13. Prior allogeneic stem cell or solid organ transplantation.
14. History of malignancy within 5 years prior to initiation of study treatment, with the exception of the cancer under investigation in this study and malignancies with a negligible risk of metastasis or death (e.g., 5-year OS (overall survival) rate > 90%) treated with an expected curative outcome, such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer.
15. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
16. Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina.
17. Major surgical procedure within 28 days prior to initiation of study treatment or anticipation of need for a major surgical procedure during the course of the study. For patients undergoing laparoscopy (without resection) for PDAC, within 14 days prior to initiation of study treatment.
18. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug or device, may affect the interpretation of the results, or may render the patient at high risk from treatment complications.
19. History of any psychiatric condition that might impair patient's ability to understand or comply with the requirements of the study or to provide consent.
20. Concurrent anti-tumor therapy beyond gemcitabine and nab-paclitaxel.
21. Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4 (cytotoxic T lymphocyte antigen-4), anti PD-1 (programmed cell death protein 1), and anti PD-L1 (programmed death-ligand 1) therapeutic antibodies.
22. Treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin 2) within 4 weeks or 5 half-lives of the drug, whichever is longer, prior to initiation of study treatment.
23. Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti - tumor necrosis factor-α [TNF-α] agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

    * Patients who received acute, low-dose, systemic immunosuppressant medications or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast-agent allergy) are eligible for the study. It is recommended that patients requiring use of steroids for a contrast-agent allergy will undergo chest CT without contrast-agent and abdomen and pelvis MRI (Magnetic Resonance Imaging) with Gadolinium.
    * Patients who received mineralocorticoids (e.g., fludrocortisone), inhaled or low-dose corticosteroids for COPD (chronic obstructive pulmonary disease) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
24. Treatment with any other investigational agent or participation in another clinical study with therapeutic intent within 28 days prior to initiation of study treatment.
25. Implantable electronic medical devices in the torso, such as pacemakers.
26. Known allergies to medical adhesives or hydrogel, or to one of the chemotherapies used in this study or biopharmaceuticals produced in Chinese hamster ovary cell products or to any component of the atezolizumab formulation.
27. Treatment with therapeutic oral or IV (intravenous) antibiotics within 2 weeks prior to initiation of study treatment.

    Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
28. Pregnant or breast-feeding, or intending to become pregnant during study treatment or within 5 months after the final dose of atezolizumab or within 6 months after the last dose of gemcitabine or within 6 months after the last dose of nab-paclitaxel, whichever is later.
29. Unable to follow the protocol for medical, psychological, familial, geographic or other reasons.
30. Admitted to an institution by administrative or court order.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2025-11-27 (Estimated); Study Completion 2025-11-27 (Estimated)

PRIMARY OUTCOMES:
Disease control rate (DCR) | at least 16 weeks for SD or confirmed PR/CR
  Disease control rate (DCR) will be measured by the proportion of patients who had either stable disease (SD) for at least 16 weeks or confirmed partial response (PR) or complete response (CR) according to RECIST v1.1

SECONDARY OUTCOMES:
Overall survival (OS) | up to 4 years
  Overall survival (OS) will be measured from time of treatment initiation until date of death.
Progression-free survival (PFS) | up to 4 years
  Progression-free survival (PFS) will be measured as the time from treatment initiation until progression per RECIST v1.1 or death.
1-Year survival rate | alive at 1 year following treatment initiation
  1 year survival rate will be measured as the percentage of patients who are alive at one year following treatment initiation .
Objective response rate (ORR) | up to 4 years
  Objective response rate (ORR) will be measured by the proportion of patients who had either complete response or partial response per RECIST v1.1 following treatment initiation.
Progression free survival at 6 months (PFS6) | 6 months following treatment initiation
  Progression free survival at 6 months (PFS6) will be measured as the proportion of patients who are not progressive per RECIST v1.1 at 6 months following treatment initiation.
Duration of response (DOR) | up to 4 years
  Duration of response (DOR) will be defined as the time from the first occurrence of a documented objective response (complete or partial response) to disease progression or death from any cause (whichever occurs first) as determined by the investigator according to RECIST v1.1.
Rate of of patients with treatment emergent adverse events | up to 4 years
  Adverse Events will be reported as incidence by body system and MedDRA term out of the number of patients who receive at least 1 day of TTFieldstreatment or one dose of atezolizumab. Based on Common Terminology Criteria for Adverse Events, CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (15):
- Czechia (4):
  - University Hospital Hradec Kralove, Hradec Králové
  - University Hospital Olomouc, Olomouc
  - University Hospital Motol, Prague
  - University Hospital Bulovka, Prague
- Germany (3):
  - Asklepios Hospital Altona, Hamburg
  - University Hospital Tuebingen, Tübingen
  - University Hospital Ulm, Ulm
- Spain (6):
  - University Hospital Vall d'Hebron, Barcelona
  - University General Hospital Gregorio Maranon, Madrid
  - University Hospital Foundation Jimenez Diaz, Madrid
  - Clara Campal Comprehensive Cancer Center (CIOCC), Madrid
  - Regional University Hospital of Malaga, Málaga
  - University Clinic of Navarra - Pamplona, Pamplona
- Switzerland (2):
  - Inselspital, University Hospital Bern, Bern
  - Fribourg Cantonal Hospital, Internal Medicine and Oncology, Fribourg

IPD SHARING:
Plan to Share IPD: No